CLINICAL TRIAL: NCT07145567
Title: Microangiopathy IN Diabetes
Acronym: MIND
Status: Recruiting | Type: Observational
Sponsor: Karolinska Institutet (Other)
Collaborators: Neko Health AB (Unknown)
Responsible Party: Principal Investigator, Sara Tehrani, Principal investigator, Medical doctor, Specialist in internal medicine, Karolinska Institutet
Other Study IDs: 2023-02232-01
Record Dates: First submitted 2025-08-21; First posted 2025-08-28 (Actual); Last update posted 2025-08-28 (Actual); Status verified 2025-02

CONDITIONS: Microangiopathy; Microvascular Complications
Keywords: Laser speckle contrast imaging; Spatial frequency domain imaging; Laser doppler flowmetry; Iontophoresis; Local thermal hyperemia; Post occlusive reactive hyperemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (4):
- Severe diabetic microangiopathy: Severe micro-angiopathy defined as proliferative retinopathy, macroalbuminuria, and kidney failure with at least CKD-class 3B and severe neuropathy with or without foot ulcers. Aged 18-60 years old.
- Moderate diabetic microangiopathy: Moderate non-proliferative retinopathy or proliferative retinopathy, macroalbuminuria or kidney failure defined as estimated glomerular filtration rate <60 mL/min/1.73 m2 body surface, and manifest neuropathy. Aged 18-45 years old.
- Mild diabetic microangiopathy: Mild-moderate non-proliferative retinopathy and/or microalbuminuria and/or early signs of neuropathy. Aged 18-45 years old.
- No diabetic microangiopathy: No microangiopathic complications, except for simplex or background retinopathy, which is an early and reversible state. Aged 18-45 years old.

SUMMARY:
This clinical trial aims to evaluate the use of a contactless and non-invasive technique to measure the properties of the skin's microcirculation and its regulatory functions in both healthy individuals and patients with microvascular disease associated with type 1 diabetes. It is hoped that the study results will lead to the development of a useful method for detecting diabetic complications at an early stage, thereby enabling treatment and preventive measures before the onset of severe microangiopathy.

DETAILED DESCRIPTION:
This study will employ investigational devices to evaluate microvascular function and correlate it to degree of microangiopathy in persons with diabetes type 1 and healthy controls.

The investigational device, TCI P4, is a novel, contactless, non-invasive, non-CE marked, class IIa Spatial Frequency Domain Imaging (SFDI) system. The device utilizes an LED light projector to cast patterned, multi-wavelength light onto the skin while multiple cameras capture narrow-band reflections. This method yields two-dimensional data on skin structure and molecular composition (including hemoglobin, oxygen, and water). Established comparators such as laser speckle contrast imaging (LSCI) and the EPOS system are employed to benchmark device performance and validate measurements.

ELIGIBILITY:
Inclusion Criteria:

* Diabetes mellitus type 1.
* Cohort specific inclusion criteria apply, please review 'groups' section.

Exclusion Criteria:

* Patients unable to understand patient information due to cognitive impairment.
* Patients unable to understand patient information due to language barriers.
* Ongoing acute infection disease or inflammatory condition.
* Pregnant or breast-feeding women.
* Patients with damaged and/or scarred tissue in the areas of interest for the investigational or comparator devices.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Outpatient at Danderyd Hospital Diabetes Clinic
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2024-03-01 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Peak perfusion in response to local thermal hyperemia | Investigation will take within 1 day from enrollment.
  As measured with investigational devices TCI P4, Pericam LSCI and EPOS devices.

SECONDARY OUTCOMES:
Perfusion heterogeneity in sole of feet | Investigation will take place within 1 day from enrollment.
  Perfusion heterogeneity index as measured by investigational device TCI P4. It will be stated as a numerical ordinal scale.

CONTACTS AND LOCATIONS:
Locations (1):
- Danderyd University Hospital, Danderyd, Stockholm County, Sweden

IPD SHARING:
Plan to Share IPD: No